CLINICAL TRIAL: NCT06914622
Title: Real-Time Experiences, Physical Activity And Biological Outcomes In Personal Recovery Of Residents With Mental Disorders (EMPOWER-RES): A Non-Randomized Multicentric Clinical Trial
Brief Title: Real-time Experiences, Physical Activity and Biological Outcomes in Personal Recovery Residents (EMPOWER-RES)
Acronym: EMPOWER-RES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Alessandra Martinelli, MD PhD Psychiatrist and clinical researcher, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0012699/25
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Severe Mental Disorder; Severe Mental Illness
Keywords: mental health supported accommodation; personal recovery; severe mental disorder; bio-psychosocial; rehabilitation
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: The study design is a non-randomized clinical trial. A group of residents receiving personal recovery-oriented treatment (N=36) will be compared to a matched group of residents receiving standard treatment (N=36). Residents in the recovery-oriented treatment group are those whose key professionals have completed specific training on personal recovery. Residents will be matched by gender, age range, and DSM-5-TR diagnostic group. Regardless of the number of residents recruited in each diagnostic category, all matched residents will be included, as their placement in the same type of supported accommodation ensures comparability in functioning and care needs. Bio-psychosocial assessments of residents, their key professionals, and informal caregivers will be conducted at baseline and at two follow-up time points: six months and nine months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recovery-oriented treatment (Experimental): A group of residents will receive a personal recovery-oriented treatment (N=36) whose key professionals have participated in specific training on personal recovery.
  Interventions: Behavioral: Mental Health Recovery Star (MHRS)
- Standard treatment (No Intervention): A group of residents will receive standard treatment (N=36). Standard residential treatment for individuals with mental disorders includes medical, psychological, and social interventions aimed at improving symptoms, quality of life, and functioning. The approach is personalized based on the individual's diagnosis, symptoms, and community resources.
  Most SAs offer personalized care plans, designated key professionals, regular individual and group activities, medication management support, and healthy lifestyle promotion. However, few facilities provide continuous psychological, vocational, and social support, adequately addressing patients' real needs.

INTERVENTIONS:
Behavioral: Mental Health Recovery Star (MHRS) — The personal recovery-oriented treatment is the Mental Health Recovery Star (MHRS), a recovery-oriented tool developed in England to support and monitor personal recovery. It features a 10-point star representing life dimensions grouped into four areas: health, functioning, self-image, and social networks. Residents assess their progress on each point using a "Scale of Change " with five recovery stages, from feeling stuck to self-reliance.
  After assessment, residents and professionals set recovery goals (up to three at a time) and create a shared care plan.
  The MHRS shows good psychometric properties, with strong validity, consistency, and ease of use, despite some inter-rater reliability issues. It is best suited for shared rehabilitation plans rather than clinical monitoring.
  Peer review meetings will be provided. The personal recovery-oriented treatment will last six months and will be considered complete upon follow-up evaluation.
  Arms: Recovery-oriented treatment

SUMMARY:
The project focuses on patients with severe mental disorders (SMD) residing in Italian mental health supported accommodation (SA). Although the goal of SA is to promote personal recovery - that is, living life to the fullest of one's potential - international literature on this topic is scarce, and traditional treatments in the Italian residential system show limitations in adopting such approaches.

The research hypothesis is that activating personal recovery pathways could improve the biopsychosocial outcomes of patients, caregivers, and professionals. To test this hypothesis, a non-pharmacological, non-randomized interventional trial will compare two groups: one group of individuals with SMD receiving recovery-oriented treatment, using the Mental Health Recovery Star, and another group of individuals with SMD receiving standard treatment.

The Mental Health Recovery Star is a ten-pointed star-shaped tool that represents various life dimensions. Patients, together with their key professional, are expected to negotiate a score for each domain on the five-stage 'Scale of Change,' capturing and monitoring the different phases of the recovery process.

DETAILED DESCRIPTION:
Interventional Study Design Primary Purpose Treatment: A personal recovery-oriented intervention is being evaluated for treating people with severe mental disorders living in mental health supported accommodations Study Phase

The project will last three years and will follow these phases:

* Phase 1: Ethical committee approval, development of the assessment manual, and training sessions for professionals. Preparation of entry and exit questionnaires for clinical and biological data collection. Establishing procedures for biological sample preparation, storage, and shipment. Conducting focus groups with patients to develop ESM questions. Setting up digital platforms and acquiring necessary materials and software. (0-8 months)
* Phase 2: Recruitment of patients, professionals, and informal caregivers at participating centers. (7-24 months)
* Phase 3: Clinical assessments and collection of biological and digital data at baseline. (7-24 months)
* Phase 4: Follow-up clinical assessments and collection of biological and digital data after six and nine months. (13-30 months)
* Phase 5: Implementation of a recovery-oriented treatment approach. (7-30 months)
* Phase 6: Supervision meetings to ensure the correct use of assessment tools. (7-30 months)
* Phase 7: Preliminary reports on interim findings, including sample description, correlation between personal recovery data and clinical variables, and initial analysis of biological and digital data. (24-30 months)
* Phase 8: Data analysis and dissemination of results through conferences, workshops, and publications. (24-36 months) Interventional Study Model Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study Model Description A group of residents receiving a personal recovery-oriented treatment (N=36) will be compared to a matched group of residents receiving standard treatment (N=36). Patients in the recovery-oriented treatment group will be those whose assigned professionals have completed specific training on personal recovery.

Patients will be matched based on sex, age range (e.g., 18-25, 26-40, 41-60, 61-70), and diagnostic group according to the DSM-5-TR (schizophrenia spectrum disorders, mood disorders, personality disorders, other). Regardless of the number of patients recruited for each diagnostic category, all patients will be included in the sample, as literature indicates that residing in a specific type of residential facility makes them comparable in terms of functioning and care needs.

Assessments will be conducted at baseline (BL) and at two follow-up time points: six months and nine months (FU).

Number of Arms Two arms. Masking No masking Allocation Nonrandomized: Participants are expressly assigned to intervention groups through a non-random method, such as those whose assigned professionals have completed or not a specific training on personal recovery.

Enrollment 72 participants: 36 for the experimental group and 36 for the control group.

ELIGIBILITY:
The study population will include:

Patients with a mental disorder inclusion criteria:

* diagnosis of a mental disorder according to DSM5TR,
* receiving treatment at an SRP of the recruiting centers,
* over 18 years old, willing to participate exclusion criteria:
* moderate/severe intellectual disability,
* inability to speak and write in Italian.

Informal caregivers of patients inclusion criteria:

* over 18 years old,
* willing to participate, exclusion criteria:
* inability to speak and write in Italian.

Mental health professionals inclusion criteria:

* working in SRPs of the recruiting centers as a psychiatrist, educator, nurse, social worker, OSS, ASA, or TeRP,
* if part of the "personal recovery-oriented treatment" group, having specific training, exclusion criteria:
* unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychosocial functioning | at baseline and at 6 and 9 months follow-up
  Personal and Social Functioning Scale (FPS): assesses four key domains (socially useful activities, personal and social relationships, self-care and hygiene, and disruptive/aggressive behaviors) with scores ranging from 0 to 100, where higher scores indicate better functioning.

SECONDARY OUTCOMES:
Rehabilitation goals | at baseline and at 6-9 months follow-up
  Valutazione delle Attività e Definizione degli Obiettivi (VADO) [Assessment of Activities and Goal Setting]: Includes the Rehabilitation Areas Module (28 items, rated on a 4-point Likert scale), where higher scores indicate higher professional interventions.
Stress-related parameters | at baseline and at 6-9 months follow-up
  Biological changes related to stress will be assessed through the collection of saliva samples (for three consecutive days) and blood samples to investigate High-sensitivity CRP, and pro-inflammatory cytokines IL-6, TNF-alpha, IL-1, IL-4, IL-10, hormone panel (Testosterone, E2, FSH, LH, SHBG, P4, PRL), concentration and size of extracellular vesicles (EVs).
Real-time experiences | at baseline and at 6-9 months follow-up for 1 week, and partly for 6 months along the experimental or control treatment
  A focus group with the patients will be conducted to collaboratively define the questions for the Experience Sampling Method (ESM) questionnaire about psychopathology, involvement in productive activities, diet, use of social media, and interpersonal relationships. Data will be explored ecologically, in real-time, and longitudinally through a custom-designed app for the project, which will send daily notifications with a brief questionnaire to be developed and administered to patients via mobile app.
Physical Activity-Related Parameters | for 1 week at baseline and at 6-9 months follow-up
  Changes in physical activity will be assessed using an accelerometer (worn for one week)
Working alliance | at baseline and at 6-9 months follow-up
  The working alliance between patients and mental health professionals will be assessed using the Working Alliance Scale (WAI 41) at BL and FU.
Psychopathology | at baseline and at 6-9 months follow-up
  Brief Psychiatric Rating Scale (BPRS): Evaluates psychopathology severity through 24 items rated on a 7-point Likert scale, covering five symptom categories (depression/anxiety, excitement, positive symptoms, negative symptoms, and cognitive symptoms). Higher scores indicate greater symptom severity.
Psychipathology and fucntioning in residential facility | at baseline and at 6-9 months follow-up
  Health of the Nation Outcome Scale - Residential Facility (HoNOS-RF): Measures personal and interpersonal functioning, environment, medical aspects, cognitive problems, and psychiatric symptoms. The 33 items are rated on a 0-4 Likert scale (higher scores indicate greater severity).
Needs for care | at baseline and at 6-9 months follow-up
  Camberwell Assessment of Need (CAN): Evaluates needs for care through a 22-item interview for both staff (CAN-S) and patients (CAN-P), rated on a 3-point scale (0 = no problem, 1 = problem managed with intervention, 2 = unmet need).
Functional autonomy in residential facility | at baseline and at 6-9 months follow-up
  Monitoring of Pathway of Rehabilitation (MPR): Assesses functional autonomy across 10 skill areas (self-care, living space maintenance, nutrition, orientation/movement, other autonomies, social skills, socio-recreational abilities, occupational skills, health management). Scores range from 0 to 12, with higher scores indicating greater functional autonomy.
Personal recovery -short | at baseline and at 6-9 months follow-up
  Hope, Agency and Opportunity (HAO): A 4-item questionnaire monitoring personal recovery, with higher scores indicating more favorable recovery outcomes.
Personal recovery | at baseline and at 6-9 months follow-up
  Recovery Assessment Scale - Domains and Stages (RAS-DS): Measures personal recovery through four key areas (hope and optimism, sense of belonging and social support, life goals and future orientation, illness management and coping skills) and five stages reflecting progress in the recovery process.
Quality of life and exploitation | at baseline and at 6-9 months follow-up
  Manchester Short Assessment of Quality of Life (MANSA): explores the patient's perception about its living situation and health. Higher scores reflect better quality of life.
Perceived functioning/disability | at baseline and at 6-9 months follow-up
  WHO Disability Assessment Schedule (WHODAS 2.0): Evaluates perceived functioning through a 12-item scale rated on a 5-point Likert scale, with higher scores indicating greater disability.
Stigma | at baseline and at 6-9 months follow-up
  Discrimination and Stigma Scale - Ultra Short (DISC-US): Measures perceived stigma through an 11-item questionnaire rated on a 4-point Likert scale, where higher scores indicate greater perceived discrimination.
Perceived loneliness | at baseline and at 6-9 months follow-up
  UCLA Loneliness Scale: A 20-item scale measuring perceived loneliness, rated on a 4-point Likert scale, with higher scores indicating greater loneliness.
Therapeutic alliance | at baseline and at 6-9 months follow-up
  Working Alliance Inventory - Short Form (WAI): Assesses therapeutic alliance using 12 items rated on a 7-point Likert scale, where higher scores indicate a stronger alliance.
Service satisfaction | at baseline and at 6-9 months follow-up
  Verona Service Satisfaction Scale - Residential Facilities (VSSS-RF): Measures service satisfaction from the patient's and informal caregiver perspective using a 24-item questionnaire rated on a 5-point Likert scale, covering overall satisfaction, staff competence, intervention effectiveness, information, access, and family involvement.
Burnout Assessment Tool (BAT) | at baseline and at 6- 9 months follow-up
  Burnout Assessment Tool (BAT): The BAT is a psychometrically valid tool, recently developed and not subject to a paid license, making it more accessible for non-profit multicenter studies.
Perceived stress | at baseline and at 6-9 months follow-up
  Perceived Stress Scale (PSS): A 10-item self-report questionnaire measuring perceived stress over the last 30 days.
Job satisfaction | at baseline and at 6-9 months follow-up
  Ad-hoc questionnaire: Evaluates job satisfaction. 11 items. higher scores indicate greater job satisfaction.
Distress | at baseline and at 6-9months follow-up
  Patient Health Questionnaire-4 (PHQ-4): A 4-item screening tool for anxiety and depression symptoms, with higher scores indicating greater distress and functional impairment.
Experiences of caregiving | at baseline and at 6-9 months follow-up
  Positive Aspects of Caregiving (PAC): Measures the positive experiences and benefits of caregiving, including feelings of usefulness, appreciation, and meaning in the caregiving relationship.
Circadian rythm- related parameters | one week at baseline and at 6-9 months follow-up
  Changes in circadian rythm will be assessed using an accelerometer
Specific Levels of Functioning Scale (SLOF) | at baseline and at 6 and 9 months follow-up
  Specific Levels of Functioning Scale (SLOF): Assesses psychosocial functioning. It consists of 43 items rated on a 5-point Likert scale, with total scores ranging from 43 to 215, where higher scores indicate better psychosocial functioning.
Triadic Interaction, aAliance, and Dynamic evaluation (TRIADE) | at baseline and at 6 and 9 months follow-up
  Triadic Interaction, aAliance, and Dynamic evaluation (TRIADE): tool for assessing the alliance and reciprocal influence within the triadic care system (25 items, 1-7 likert scale; higher scores indicate stronger influence; validation ongoing)
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | at baseline and at 6-9 months follow-up
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS):
  Assesses cognitive functions through 12 subtests grouped into 5 index scores. Scores below the mean indicate cognitive difficulties or possible impairment.
Resilience Scale - 14 item (RS-14): | at baseline and at 6 and 9 months follow-up
  Resilience Scale - 14 item (RS-14): Measures personal resilience across 14 items; higher scores indicate greater resilience.
Quality Indicator for Rehabilitative Care - Short Assessment (QuIRC-SA) | once in 6 months from the baseline
WHO Quality of Life-Brief scale (WHOQOL-Brief) | at baseline and at 6 and 9 months follow-up
  WHO Quality of Life-Brief scale (WHOQOL-Brief): Assesses quality of life (26 items, 4 domains, 5-point Likert scale, range 0-100; higher scores indicate better quality of life).
Zarit Burden Interview (ZBI) | at baseline and at 6 and 9 months follow-up
  Zarit Burden Interview (ZBI): Measures caregiver burden (29 items, 6 domains, 0-4 Likert scale; higher scores indicate greater burden).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Martinelli, MD PhD, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy
Locations (3):
- Italy (3):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Centro Sacro Cuore di Gesù, San Colombano al Lambro (MI), Milan
  - Centro Sant'Ambrogio, Cernusco sul Naviglio (MI), Milan

IPD SHARING:
Plan to Share IPD: Yes
To promote open, transparent, and collaborative science, the raw data from all studies conducted at the IRCCS Fatebenefratelli will be published in publicly accessible repositories, as required by the scientific community and funding bodies, including the Ministry of Health and the European Commission. The raw clinical and biological data related to participants in this research, a non-randomized multicenter non-pharmacological clinical trial, will be published in a form that ensures the protection of participants' privacy in accordance with current regulations. Repositories will be selected that allow access to the information only after authentication of the access request and validation by the study responsible (or a designated representative) of the reasons for the request. The public repository will also be chosen based on the cybersecurity and data protection guarantees it offers.
Supporting Information: Study Protocol
Time Frame: From December 2028 to Dcember 2029
Access Criteria: De-identified clinical and biological data from this non-randomized multicenter trial will be available in secure public repositories to support open science.
  * Eligibility: Access is granted for research aligned with study objectives, including secondary and meta-analyses. Requests must detail statistical methods, subject to independent review.
  * Privacy & Security: Data will comply with protection regulations, stored only in repositories with strong cybersecurity measures.
  * Access Process: Researchers must submit a formal request and sign a Data Sharing Agreement (DSA) before access is granted. Authentication via the repository's system is required.
  * Review & Approval: Requests will be evaluated by the study lead (or representative) based on scientific merit, ethical compliance, and feasibility.